CLINICAL TRIAL: NCT01023906
Title: Relationship Between Variations in Taste Perception and Chronic Disease Risk Factors as a Function of Age
Brief Title: Taste Perception and Chronic Disease Risk
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Sponsor
Other Study IDs: Ross Aging Initiative
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Cardiovascular Disease; Diabetes; Obesity; Metabolic Syndrome; Aging
Keywords: Taste; general Labeled Magnitude Scale; Aging; Chronic Disease Risk; Smell
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Obesity; Metabolic Syndrome; Anosmia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood, and DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 18-49 years: Younger
- 50-85 years: Older

SUMMARY:
The purpose of the Taste Perception Study is to assess variations in the ability to taste and perceive sensations from various stimuli in younger (18-49 years) and older (50-85 years) volunteers. The study's goal is to determine how these sensations influence what one likes to eat, and what one chooses to eat, and whether there is an association with dietary intake, body composition and chronic disease. Another objective of the study is to determine the association between variations in oral sensations and genes mediating sensory perception and dietary behaviours.

DETAILED DESCRIPTION:
The objective of the Taste Perception Study is to assess variations in oral sensations in younger (18-49 years; n=35) relative to older (50-85 years; n=35) subjects, and determine the association between variations in oral sensations and measures of chronic disease risk factors, body composition, habitual dietary intake and selected genes mediating sensory perception and dietary behaviors. Subjects who are participating in the Glycemic Index study (IRB #7196) will be asked for voluntarily participation in the proposed study. These volunteers will undergo 1-2 hours of standardized testing. These tests will involve tasting or smelling certain foods/beverages or ingredients in foods/beverages and rating the degree of liking/disliking, intensity and flavor or odor using a validated general Labeled magnitude scale. Volunteers will also be asked to complete a food preference survey and eating inventory questionnaire, as well as provide a DNA sample from a cheek swab or blood sample. These data will then be merged with the measures of chronic disease risk factors, body composition and habitual dietary intake data generated from the Glycemic index study in order to better understand if variations in oral sensations influence food preferences and patterns and subsequently chronic disease risk.

ELIGIBILITY:
Inclusion Criteria:

* men and women;
* aged 18 to 85 years old;
* free of known chronic disease;
* BMI < 35 kg/ m2.

Exclusion criteria:

* BMI ≥ 35 kg/m2;
* renal or liver disease;
* untreated hypertension;
* irritable bowel syndrome;
* malabsorptive, esophageal and gastrointestinal motility disorders;
* chronic pancreatitis, or history of acute pancreatitis within the last year;
* hypothyroidism or hypothyroidism, as defined as screening TSH outside of normal ranges;
* anemia, as defined by screening hematocrit of 34% for women and 38% for men;
* smoking within the past 6 months;
* diabetes;
* fasting glucose ≥ 125 mg/dL;
* pregnancy or breastfeeding;
* history of polycystic ovary syndrome;
* history of autoimmune or other connective tissue disorders associated with chronic inflammation, such as rheumatoid arthritis; alcohol consumption > 7 drinks/ week;
* use of medications known to affect glucose or lipid metabolism;
* established CVD (myocardial infarction, stroke, heart failure, coronary artery bypass, graft, stenosis > 50%, peripheral arterial disease);
* unwillingness to adhere to study protocol;
* weight gain or loss of more than 15 lbs within 6 months prior to enrollment and other abnormal screening laboratory analysis results.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Sensory/hedonic rating | 1 - 2 hours

SECONDARY OUTCOMES:
Genetic Variation | 1- 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nirupa R Matthan, Ph.D., Principal Investigator — HNRCA at Tufts University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Vega-Lopez S, Ausman LM, Griffith JL, Lichtenstein AH. Interindividual variability and intra-individual reproducibility of glycemic index values for commercial white bread. Diabetes Care. 2007 Jun;30(6):1412-7. doi: 10.2337/dc06-1598. Epub 2007 Mar 23. PMID 17384339
- [Background] He W, Sengupta M, Velkoff VA, DeBarros KA. U.S. Census Bureau, Current Population Reports, 65+ in the United States: 2005. U.S. Government Printing Office, Washington DC. 2005: 23-209.
- [Background] Duffy VB, Chapo AK. Smell, Taste, and Somatosensation in the Elderly. Jones and Bartlett Publishers, 2006: 115-153.
- [Background] Seiberling KA, Conley DB. Aging and olfactory and taste function. Otolaryngol Clin North Am. 2004 Dec;37(6):1209-28, vii. doi: 10.1016/j.otc.2004.06.006. PMID 15563911
- [Background] Dinehart ME, Hayes JE, Bartoshuk LM, Lanier SL, Duffy VB. Bitter taste markers explain variability in vegetable sweetness, bitterness, and intake. Physiol Behav. 2006 Feb 28;87(2):304-13. doi: 10.1016/j.physbeh.2005.10.018. Epub 2005 Dec 20. PMID 16368118
- [Background] Bartoshuk LM, Duffy VB, Hayes JE, Moskowitz HR, Snyder DJ. Psychophysics of sweet and fat perception in obesity: problems, solutions and new perspectives. Philos Trans R Soc Lond B Biol Sci. 2006 Jul 29;361(1471):1137-48. doi: 10.1098/rstb.2006.1853. PMID 16815797
- [Background] Drewnowski A. Taste preferences and food intake. Annu Rev Nutr. 1997;17:237-53. doi: 10.1146/annurev.nutr.17.1.237. PMID 9240927
- [Background] Lanier SA, Hayes JE, Duffy VB. Sweet and bitter tastes of alcoholic beverages mediate alcohol intake in of-age undergraduates. Physiol Behav. 2005 Jan 17;83(5):821-31. doi: 10.1016/j.physbeh.2004.10.004. Epub 2004 Nov 21. PMID 15639168
- [Background] Goldstein GL, Daun H, Tepper BJ. Adiposity in middle-aged women is associated with genetic taste blindness to 6-n-propylthiouracil. Obes Res. 2005 Jun;13(6):1017-23. doi: 10.1038/oby.2005.119. PMID 15976144
- [Background] Duffy VB. Associations between oral sensation, dietary behaviors and risk of cardiovascular disease (CVD). Appetite. 2004 Aug;43(1):5-9. doi: 10.1016/j.appet.2004.02.007. PMID 15262011
- [Background] Rolls BJ. Do chemosensory changes influence food intake in the elderly? Physiol Behav. 1999 Apr;66(2):193-7. doi: 10.1016/s0031-9384(98)00264-9. PMID 10336143
- [Background] Bartoshuk LM, Duffy VB, Miller IJ. PTC/PROP tasting: anatomy, psychophysics, and sex effects. Physiol Behav. 1994 Dec;56(6):1165-71. doi: 10.1016/0031-9384(94)90361-1. PMID 7878086
- [Background] Bartoshuk LM, Duffy VB, Fast K, Green BG, Prutkin K, Snyder DJ. Labeled scales (e.g. category, Likert, VAS) and across-group comparisons: what we have learned from genetic variation in taste. Food Quality and Preference 2003; 14: 125-138.
- [Background] Green BG, Dalton P, Cowart B, Shaffer G, Rankin K, Higgins J. Evaluating the 'Labeled Magnitude Scale' for measuring sensations of taste and smell. Chem Senses. 1996 Jun;21(3):323-34. doi: 10.1093/chemse/21.3.323. PMID 8670711